CLINICAL TRIAL: NCT05822609
Title: Trial of Semaglutide for Diabetic Kidney Disease in Type 1 Diabetes
Acronym: RT1D
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of Colorado, Denver (Other); Providence Healthcare (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Ian deBoer, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00016349
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Kidney Disease; Type 1 Diabetes
Keywords: Glucagon-like peptide-1 receptor agonist
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide group from 0.25mg to 1.0mg
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Semaglutide — 1.0 mg
  Arms: Semaglutide
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effects of semaglutide on kidney oxygenation and function in type 1 diabetes. The secondary objective is to determine the glycemic effects and safety of semaglutide in type 1 diabetes.

DETAILED DESCRIPTION:
A parallel-group, double-blind, placebo-controlled, randomized study will rigorously test effects of semaglutide on the kidney. Real-time continuous glucose monitoring will be used to control glycemia during study run-in (prior to randomization) and during active therapy, which investigators anticipate will lead to similar glycemic control according to treatment assignment and ability to assess effects independent of glycemia. The trial duration is 26 weeks, a period of time sufficient to gradually titrate study medications to maximum target dose (over 12 weeks) and then observe the full short-term effect of semaglutide on the kidney.

Study Aims and Hypotheses:

Aim 1: Determine the effects of semaglutide vs. placebo on kidney oxygenation in type 1 diabetes. Hypothesis 1: Semaglutide will improve kidney oxygen availability in adults with type 1 diabetes.

Aim 2: Determine the effects of semaglutide vs. placebo on urine albumin-creatinine ratio and estimated glomerular filtration rate in type 1 diabetes. Hypothesis 2: Semaglutide will lower albuminuria and slow estimated glomerular filtration rate decline in adults with type 1 diabetes.

Aim 3: Determine the glycemic effects and safety of semaglutide vs. placebo in type 1 diabetes. Hypothesis 3: Semaglutide will reduce total daily insulin dose and improve glycemic variability without increasing risk of severe hypoglycemia or diabetic ketoacidosis in adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with type 1 diabetes
* Diabetes duration of ≥5 years
* Persistent urine albumin-to-creatinine ratio (UACR) ≥ 30 mg/g, on the most recent two measurements within the prior 3 years
* Estimated glomerular filtration rate ≥ 30 mL/min/1.73m2
* Stable doses of drugs altering blood pressure (e.g., Angiotensin-converting enzyme inhibitor) required for at least 4 weeks prior to randomization, and requested for the duration of the trial
* Stable doses of lipid-lowering medications required for at least 4 weeks prior to randomization, and requested for the duration of the trial
* Adequate contraceptive method for females of child-bearing potential

Exclusion Criteria:

* HbA1c >9%, recent diabetic ketoacidosis, hyperosmolar hyperglycemic state or severe illness requiring hospitalization in past 30 days
* Other causes of diabetes mellitus, including type 2 diabetes and maturity-onset diabetes of the young (MODY)
* Chronic kidney disease unrelated to diabetes
* Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2) or thyroid nodule palpated by endocrinologist at screening
* Personal history of pancreatitis
* Current/planned pregnancy or nursing
* Uncontrolled thyroid disease or hypertension (Systolic blood pressure [SBP] ≥ 160 mm Hg or diastolic blood pressure [DBP] ≥ 100 mm Hg despite treatment)
* Proliferative retinopathy with treatment in the past 6 months
* Uncontrolled or potentially unstable diabetic retinopathy or maculopathy, verified by fundus examination with pupil dilation unless performed using a digital fundus photography camera specified for non-dilated examination
* More than 2 severe hypoglycemic episodes (requiring glucagon and/or assistance from another person) in the past 6 months
* Frequent hypoglycemia during the last two weeks of the study run-in phase (time below range [<70 mg/dL] ≥4%)
* Pramlintide and the use of glycemia treatments not approved for type 1 diabetes by the FDA, e.g., metformin, SGT-2 inhibitor, GLP-1 receptor agonist, closed loop insulin delivery using unapproved algorithms
* Significant systemic conditions or treatment such as cancer or immunomodulators
* Known liver disease other than non-alcoholic fatty liver disease (NAFLD) or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >100 IU/L, history of severe gastrointestinal disease (e.g., gastroparesis) or gallstones
* Body mass index <20 kg/m2
* Inability to cooperate with or clinical contraindication for magnetic resonance imaging including severe claustrophobia, nonremovable devices, implanted metal
* Known or suspected allergy/sensitivity to semaglutide or its excipients
* Pregnant, breast feeding, or the intention of becoming pregnant
* The receipt of any investigational drug within 3 months prior to this trial
* Previously randomized in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in kidney cortical relaxation rates (R2*) | Baseline to 26 weeks
  Measurement of oxygenation by magnetic resonance imaging

SECONDARY OUTCOMES:
Change in urine albumin excretion | Baseline to 26 weeks
  Measured as mean of multiple urine albumin-creatinine ratio measurements in spot urine
Change in estimated glomerular filtration rate | Baseline to 26 weeks
  Estimated glomerular filtration rate will be calculated from age, sex, and the serum concentrations of creatinine and cystatin C
Change in glucose time in range | Baseline to 26 weeks
  Proportion of time with glucose 70-180 mg/dL measured by continuous glucose monitoring
Change in glucose coefficient of variation | Baseline to 26 weeks
  Measured by continuous glucose monitoring
Change in total daily insulin dose | Baseline to 26 weeks
  Mean total dose of insulin administered per day

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, MD, MS, Principal Investigator — University of Washington; Jessica Kendrick, MD, Principal Investigator — University of Colorado Anschutz Medical Campus and Children's Hospital Colorado; David Cherney, PhD, MD, Principal Investigator — University of Toronto; Irl Hirsch, MD, Principal Investigator — University of Washington; Katherine Tuttle, MD, Principal Investigator — Providence Healthcare
Locations (4):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Washington, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study team will field direct requests from other researchers to share deidentified data after completion of the trial.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Kugathasan L, Aronson Y, Sridhar VS, Ni H, Ouimet JP, Limonte CP, Sarma S, Cherney DZI. Advancing kidney protection in type 1 diabetes: insights from emerging therapies in type 2 diabetes and chronic kidney disease. Expert Rev Clin Immunol. 2025 Aug;21(8):1113-1134. doi: 10.1080/1744666X.2025.2537446. Epub 2025 Jul 24. PMID 40693871